CLINICAL TRIAL: NCT00003396
Title: Evaluation of Allogeneic Peripheral Blood Stem Cell Transplants From a Related Donor Without Graft-Versus-Host Prophylaxis in Patients With High Risk of Relapse
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000066397; MSGCC-9805; NCI-V98-1430
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute eosinophilic leukemia; adult acute basophilic leukemia; adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute promyelocytic leukemia (M3); childhood acute erythroleukemia (M6); childhood acute eosinophilic leukemia; childhood acute basophilic leukemia; childhood acute megakaryocytic leukemia (M7); recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Erythroblastic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Megakaryoblastic, Acute; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Antilymphocyte Serum; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: graft-versus-tumor induction therapy
Drug: cyclophosphamide
Drug: melphalan
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation from related donors to prevent graft-versus-host disease in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the use of donor peripheral blood stem cells without graft-versus-host disease prophylaxis to maximize the probability of graft-versus-tumor effect in patients with hematologic malignancies refractory to standard chemotherapy and unlikely to be cured with high dose chemotherapy and radiotherapy.

OUTLINE: Prior to peripheral blood stem cell transplant, patients undergo preparative cytoreduction. Patients receive total body irradiation (TBI) beginning on day -5. Radiotherapy is administered in 9 doses over 3 days (3 doses per day for 3 days). Male patients with acute lymphocytic leukemia receive an additional dose of radiation to the testicles. Patients who are ineligible for TBI due to prior radiotherapy receive 2 doses of melphalan IV on day -3. All patients receive cyclophosphamide IV over 1 hour on days -2 and -1. Anti-thymocyte globulin is also administered IV over 6 hours on days -2 and -1. Approximately 24-36 hours after the last dose of cyclophosphamide, peripheral blood stem cells obtained from the HLA matched related donor are infused into the patient. Patients do not receive graft-versus-host disease prophylaxis after transplant; however, all other forms of supportive care are provided. Patients are followed for 1 year.

PROJECTED ACCRUAL: A maximum of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients with HLA identical family donors and any one of the following conditions documented by marrow aspiration and biopsy: -Acute leukemia refractory to induction treatment or after 1 or more relapses -Acute myeloid leukemia with t(9;22), -5/5q-, -7/7q-, and 11q23 involvement in first remission (not M4 or M5) -Acute lymphocytic leukemia with t(9;22) or t(4;11) in first remission -Myelodysplastic syndrome with greater than 5% bone marrow blasts -Chronic myeloid leukemia in accelerated phase or nonlymphoid blast crisis -Myeloma, chronic lymphocytic leukemia, non-Hodgkin's lymphoma, or Hodgkin's disease refractory to 2 lines of standard treatment or progression on standard treatment No evidence of active extramedullary disease

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 70-100% Life expectancy: Greater than 8 weeks Hematopoietic: Not specified Hepatic: Bilirubin less than 2.0 mg/dL SGOT no greater than 4 times upper limit of normal and not increasing for 2-4 weeks prior to transplant Renal: Creatinine less than 2 times normal and not increasing for 2-4 weeks prior to transplant OR Creatinine clearance greater than 60 mL/min Cardiovascular: LVEF greater than 50% by MUGA Pulmonary: DLCO greater than 50% Other: Not HIV positive Not pregnant or nursing Fertile patients must use effective contraceptive

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 1998-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry R. Meisenberg, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States